CLINICAL TRIAL: NCT04514965
Title: Measuring Macrophage Activation Markers and Influence on Bile Acid Composition in Patients With Primary Biliary Cholangitis After Treatment With Bezafibrate
Brief Title: Bezafibrate in Patients With Primary Biliary Cholangitis (PBC)
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PBC Beza AU
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Bezafibrate; Macrophage activation markers; Fibrosis markers; Bile acid composition
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PBC patients offered bezafibrate treatment: All patients started on bezafibrate treatment are offered inclusion in the study.
  First visit is before start of treatment. Afterwards patients will be seen at 4 weeks, 6 months, 1 year, 2 years and 3 years after inclusion.
  At all visits blood samples will be taken and liver stiffness will be measured using FibroScan. Further, they will be asked about pruritus.
  Interventions: Other: Blood sampling; Device: Fibroscan; Other: Question

INTERVENTIONS:
Other: Blood sampling — Blood sampling
Device: Fibroscan — Measurement of liver stiffness
Other: Question — Question about pruritus

SUMMARY:
Up to 40% of patients with PBC have an inadequate response to standard treatment with UDCA, hence bezafibrate, a PPAR-agonist is being introduced as add-on therapy in these patients. sCD163, fibrosis markers and bile acid composition are of special interest in PBC. In this study, the investigators will investigate how treatment with bezafibrate influence levels of macrophage activation markers and fibrosis markers as well as bile acid composition in patients offered bezafibrate as add-on therapy to UDCA.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC) is an autoimmune cholestatic liver disease characterized by destruction of intrahepatic bile ducts and progression to liver fibrosis and cirrhosis. The diagnosis of PBC is based on the presence of two of three major criteria; unexplained serum alkaline phosphatase (ALP) >1.5 times upper normal limit for more than 24 weeks, presence of anti-mitochondrial antibodies (AMA), and compatible liver histology.

Ursodeoxycholic acid (UDCA) is currently the only approved drug used to treat PBC and patients treated with UDCA have improved survival. In Denmark all PBC patients are offered UDCA treatment. However, up to 40% of PBC patients may be classified as insufficient responders to UDCA treatment with male gender, low age, and low Vitamin D level at diagnosis associated with insufficient response. More precise predictors of insufficient response to UDCA treatment are important to find as insufficient responders have worse 10-year survival probability than responders. The high proportion of insufficient responders has fuelled the search for novel treatment options, including fibrates, budesonide, and obeticholic acid. Despite response to UDCA treatment, liver transplantation remains the only cure for PBC and patients with expected survival less than one year are potential candidates for liver transplantation.

Bezafibrate Bezafibrate is a pan-peroxisome proliferator-activated receptor (PPAR) agonist. For decades, bezafibrate has been prescribed for various indications including hyperlipidemia. Thus, adverse effects are well described. Recently, a phase 3 trial showed promising results as an add-on therapy to UDCA in reducing ALP in PBC patients, who had insufficient response to UDCA alone. Hence, Danish hepatologists are starting to use bezafibrate as second line, add-on, therapy in PBC patients.

Soluble CD163 and fibrosis markers In PBC, inflammation is attributed to an immune response to mitochondrial autoantigens followed by development of anti-mitochondrial antibodies (AMAs); and accompanied by inflammation of small bile ducts. The pathogenesis includes both CD4 and CD8 cells, which in the presence of biliary cells expressing the 2-oxo-dehydrogenase pathway (PDC-E2) activates macrophages via granulocyte macrophage colony-stimulating factor. The activated macrophages, together with AMAs, produce a proinflammatory response with subsequent liver inflammation and fibrosis. Thus, macrophages seem to be involved in PBC disease severity and progression. The investigators recently showed that the macrophage activation marker soluble (s)CD163 is associated with long-term prognosis in PBC patients. Further, the investigators research group have shown increased levels of sCD163 in relation to liver fibrosis/cirrhosis in patients with chronic viral hepatitis (HBV and HCV), non-alcoholic fatty liver disease (NAFLD/NASH) and alcoholic liver disease (alcoholic hepatitis and cirrhosis) and liver disease severity including risk of portal hypertension and development of complications and mortality. Moreover, the investigators also demonstrated sCD163 is associated with early and long-term prognosis of patients with cirrhosis and acute-on-chronic liver failure.

Fibrosis is a hallmark of liver disease progression and extracellular matrix (ECM) turnover is a prominent feature of chronic inflammatory liver diseases including PBC. ECM protein degradation and formation generate fragments reflecting aspects of the tissue turnover balance when quantified in the blood. PRO-C3 and PRO-C4 reflect type III and IV collagen formation, whereas C3M and C4M are markers for degradation of type III and IV. The investigators aim to investigate changes in these fibrosis markers before and after bezafibrate treatment, to demonstrate if these novel finger print protein biomarkers may be useful for treatment response in PBC patients.

Bile acids In PBC there is intrahepatic accumulation of potentially cytotoxic bile acids resulting in liver damage. Further the composition of bile acids is changed, resulting in changes of microbiota and in the integrity of the intestinal wall, potentially allowing an increased flux of inflammatory metabolites to the liver. Exploration of potential changes in bile acid profile caused by bezafibrate treatment may improve understanding of the treatment effects and provide identification of specific treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* PBC patient offered bezafibrate treatment

Exclusion Criteria:

* patient age under 18
* life expectancy less than 6 months
* known cancer
* planned liver transplantation within 6 months
* other liver disease (viral, autoimmune, alcohol, NAFLD/NASH)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with inadequate response to UDCA treatment (ALP>170 I/U), who are offered, and accept, add-on treatment with bezafibrate at Aarhus University hospital or Hvidovre hospital are invited to partipate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Treatment effect on sCD163 levels | 4 weeks to 3 years
  Treatment effect on sCD163 levels measured in mg/L
Treatment effect on levels of fibrosis markers | 4 weeks to 3 years
  Treatment effect on levels of fibrosis markers
Treatment effect on liver stiffness | 4 weeks to 3 years
  Treatment effect on liver stiffness measured in kilopascal
Treatment effect on bile acid composition | 4 weeks to 3 years
  investigation of bile acid composition before and after treatment

SECONDARY OUTCOMES:
Treatment effect on the degree of pruritus | 4 weeks to 3 years
  Treatment effect on the degree of pruritus measured using questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Prof, MD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Hepatology and Gastroenterology, Aarhus University Hospital, Denmark, Aarhus N, Central Jutland
  - Department of Medicine, Gastrounit Medical division, Hvidovre

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided